CLINICAL TRIAL: NCT05508815
Title: The Efficacy and Safety of the Modified Zhiwang Decoction Combined With Methotrexate in Early Rheumatoid Arthritis
Brief Title: Modified Zhiwang Decoction Combined With Methotrexate in the Treatment of Early Rheumatoid Arthritis
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, zhang liubo, MD, Beijing University of Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: zliubo
Record Dates: First submitted 2022-08-15; First posted 2022-08-19 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Zhiwang Decoction Combined with Methotrexate (Experimental)
  Interventions: Drug: Modified Zhiwang Decoction Combined with methotrexate
- Methotrexate (Active Comparator)
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Modified Zhiwang Decoction Combined with methotrexate — Modified Zhiwang Decoction 100 ml (twice, per day) and methotrexate (7.5-15mg, once a week) for 12 weeks.
  Arms: Modified Zhiwang Decoction Combined with Methotrexate
Drug: Methotrexate — Methotrexate(7.5-15mg, once a week) for 12 weeks.
  Arms: Methotrexate

SUMMARY:
The aim of this study is to evaluate the effectiveness and safety of Modified Zhiwang Decoction in combination with methotrexate for the treatment of early RA patients and a parallel-group, single-center randomized controlled clinical study was designed.

DETAILED DESCRIPTION:
Rheumatoid Arthritis(RA) is a progressive inflammatory autoimmune disease characterized by chronic systemic inflammation, which can cause swelling, stiffening and articular cartilage and bone destruction. Early diagnosis and treatment in RA can improve outcomes and slow progression of joint damage. Modified Zhiwang Decoction(MZWD) has great curative effects for treating RA. However, few randomized clinical trials(RCTs) have evaluated the effectiveness of MZWD for the treatment of early RA. Therefore, a parallel-group randomized controlled trial was designed to evaluate the efficacy and safety of MZWD combined with methotrexate on early RA.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 16-70 years old;
* Patients who meet the diagnostic criteria of 2010 ACR/EULAR .
* Patients who meet the diagnostic criteria of cold pattern.
* Disease activity score(DAS28) ≤5.2.

Exclusion Criteria:

* Patients accompanied with other rheumatic diseases or severe pain due to other medical conditions, such as diabetic pain or post-herpetic neuralgia;
* Patients with joint dysfunction and the X-ray score of wrists is grade IV;
* Patients accompanied with mental and psychological disorders such as cognitive impairment, depression, anxiety, physical dysfunction, cerebral infarction, cerebral hemorrhage, epilepsy, TIA, myelitis, demyelinating disease and other central nervous system diseases.
* Patients accompanied with organ injury or malignant tumors, disorders of the cardiovascular system, liver(ALT/AST>3 times higher than the upper limit of normal), kidneys(Ccr<60ml/min), brain, or hematopoietic system.
* Pregnant and lactating women.
* Patients are participation in any other clinical trials.
* Patients who are allergic to the drugs used in this study.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-02-09 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
DAS28 based on erythrocyte sedimentation rate scores | 12 weeks
  DAS28 is widely accepted to evaluate RA disease activity and consists of number of tender joints out of 28, number of swollen joints out of 28, ESR and the patient's global assessment of disease activity.

SECONDARY OUTCOMES:
Fatigue scale-14 | 12 weeks
  The fatigue scale-14 is a standardized questionnaire regarding physical and mental fatigue. The higher the score, the greater the fatigue.
Visual analogue scale pain scores | 12 weeks
  Visual analogue scale pain score is utilized to quantify the pain level that ranges from 0 to 10. A VAS score of 0 means no pain and a score of 10 means unbear-able pain.
Traditional chinese medicine symptom scores | 12 weeks
  Traditional chinese medicine symptom score is calculated based on the percentage of symptom score reduction(PSSR) and the formula is as follows:
  PSSR=((symptom score before treatment-symptom score after treatemt)/(symptom score before treatment))×100%
Erythrocyte sedimentation rate | 12 weeks
C-reactive protein | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Xu, Study Chair — China-Japan Friendship Hospital; Cheng Xiao, Study Director — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang N, Zhang LB, Wang Z, Lan TY, Wang JP, Xiao C, Tao QW, Xu Y. Efficacy and safety of the modified Zhiwang decoction combined with methotrexate in early rheumatoid arthritis: study protocol for a randomised controlled trial. BMJ Open. 2024 Jan 18;14(1):e076571. doi: 10.1136/bmjopen-2023-076571. PMID 38238175